CLINICAL TRIAL: NCT02364245
Title: Design and Evaluation the Feasibility, Effects of Kinect-based Computer Games as Upper Extremity Training Tool in Children With Cerebral Palsy
Brief Title: Evaluation the Feasibility and Effects of Kinect-based Computer Games as UE Training Tool in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8D0941
Record Dates: First submitted 2015-01-26; First posted 2015-02-18 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2014-11

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy.; Upper Extremity; Kinect; Virtual reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinect (Experimental): Receive computer games training for 30 minutes and 30 minutes traditional OT.There are 3 sections for 1 week; the intervention period will be 8 weeks.
  Interventions: Device: Kinect; Other: Traditional OT(30 Mins)
- Traditional (Placebo Comparator): The control group will receive traditional OT for 1 hour. There are 3 sections for 1 week; the intervention period will be 8 weeks.
  Interventions: Other: Traditional OT(60 Mins)

INTERVENTIONS:
Device: Kinect — Receive computer games training for 30 minutes. There are 3 sections for 1 week; the intervention period will be 8 weeks.
  Arms: Kinect
Other: Traditional OT(30 Mins) — Receive Traditional Occupational Therapy training for 30 minutes. There are 3 sections for 1 week; the intervention period will be 8 weeks.
  Arms: Kinect
Other: Traditional OT(60 Mins) — Receive Traditional Occupational Therapy training for 60 minutes. There are 3 sections for 1 week; the intervention period will be 8 weeks.
  Arms: Traditional

SUMMARY:
The purpose of this study is to design and evaluation the feasibility, effects of Kinect-based Computer Games as Upper Extremity Training Tool in Children with Cerebral Palsy.

DETAILED DESCRIPTION:
Background Children with cerebral palsy (CP) usually have various limitations in function of their upper limbs. Upper limbs function training is one of the important issues in CP rehabilitation. There is a growing interest in rehabilitation specialists to integrate commercialized interactive computer play into rehabilitation programs. According to the literature research, commercialized interactive computer play could improve speed and quality of movement, for hand or upper limb function, the results were mixed. The investigators think the interactive computer play could be feasible in upper limb training among children with CP. However, the investigators should integrate the rehabilitation training concept to the computer playing in order to get better outcome from such training. The electronic experts and rehabilitation experts should work together to reach the goal. Therefore, the aims of this study are 1.to design Kinect computer games as the rehabilitation training tool for upper limbs of children with CP, 2. to assess the feasibility and effects of the Kinect computer games.

Methods The investigators will spend around nine months to design the computer games. The investigators will search from the internet to download the computer games which are with no copy-right issue. The investigators will use Kinect sensor to catch the child's motion. The rehabilitation team will choose several upper limb motions which are common used in training for children with CP. Then Professor Chang's team will modify the software design to make those target motions to be the game control actions.When a prototype game is created, the investigators will invite two to four children with CP to pilot test the game. The game design will be completed till children and therapists satisfy the design.

Within one year and three months the investigators will do a randomized control trial to compare the effects between the Kinect games and traditional occupational therapy (OT) in the upper limb function of children in CP. The investigators will recruit 30 children and randomize them into two groups.

In each intervention section the intervention group will receive computer games training for 30 minutes and 30 minutes traditional OT. The control group will receive traditional OT for 1 hour. There are 3 sections for 1 week; the intervention period will be 8 weeks.

Statistic methods Inter-group differences in baseline characteristics were evaluated using an independent t tests or Wilcoxon rank sum tests or χ2 analysis. Analysis of variance with repeated measures was used to determine the effects of intervention on each dependent variable. Model effects were group, time, and their interaction.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* 4-12 years old
* Cognition ability is good for evaluation and training
* Affected side: Manual ability classification system(MACS) I-III

Exclusion Criteria:

* Accept Upper Extremity surgery before recruiting
* Accept Botox injunction three months before recruiting
* Unstable Seizure

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Melbourme Assessment Scales | Children will be assesed at 8 weeks and 16 weeks

SECONDARY OUTCOMES:
Change from Baseline in Quality of Upper Extremity Skills Test | Children will be assesed at 8 weeks and 16 weeks
Change from Baseline in Motor-free perceptual assessment | Children will be assesed at 8 weeks and 16 weeks
Change from Baseline in ABILHAND-kids | Children will be assesed at 8 weeks and 16 weeks
Change from Baseline in Box and Block Test | Children will be assesed at 8 weeks and 16 weeks
Change from Baseline in Cerebral Palsy Quality of Life for Children (CP QOL-Child) questionnaire | Children will be assesed at 8 weeks and 16 weeks
Change from Baseline in Visual analogue scale | Children will be assesed at 8 weeks and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Wen Hung, MD, Principal Investigator — Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan
Locations (1):
- Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon AM. To constrain or not to constrain, and other stories of intensive upper extremity training for children with unilateral cerebral palsy. Dev Med Child Neurol. 2011 Sep;53 Suppl 4:56-61. doi: 10.1111/j.1469-8749.2011.04066.x. PMID 21950396
- [Background] Gordon AM, Charles J, Wolf SL. Methods of constraint-induced movement therapy for children with hemiplegic cerebral palsy: development of a child-friendly intervention for improving upper-extremity function. Arch Phys Med Rehabil. 2005 Apr;86(4):837-44. doi: 10.1016/j.apmr.2004.10.008. PMID 15827942
- [Background] Gordon AM, Charles J, Wolf SL. Efficacy of constraint-induced movement therapy on involved upper-extremity use in children with hemiplegic cerebral palsy is not age-dependent. Pediatrics. 2006 Mar;117(3):e363-73. doi: 10.1542/peds.2005-1009. PMID 16510616
- [Background] Wu WC, Hung JW, Tseng CY, Huang YC. Group constraint-induced movement therapy for children with hemiplegic cerebral palsy: a pilot study. Am J Occup Ther. 2013 Mar-Apr;67(2):201-8. doi: 10.5014/ajot.2013.004374. PMID 23433275
- [Background] Taub E, Ramey SL, DeLuca S, Echols K. Efficacy of constraint-induced movement therapy for children with cerebral palsy with asymmetric motor impairment. Pediatrics. 2004 Feb;113(2):305-12. doi: 10.1542/peds.113.2.305. PMID 14754942
- [Background] Sakzewski L, Ziviani J, Abbott DF, Macdonell RA, Jackson GD, Boyd RN. Participation outcomes in a randomized trial of 2 models of upper-limb rehabilitation for children with congenital hemiplegia. Arch Phys Med Rehabil. 2011 Apr;92(4):531-9. doi: 10.1016/j.apmr.2010.11.022. PMID 21440700
- [Background] Galvin J, McDonald R, Catroppa C, Anderson V. Does intervention using virtual reality improve upper limb function in children with neurological impairment: a systematic review of the evidence. Brain Inj. 2011;25(5):435-42. doi: 10.3109/02699052.2011.558047. Epub 2011 Mar 14. PMID 21401370
- [Background] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008349. doi: 10.1002/14651858.CD008349.pub2. PMID 21901720
- [Background] Fehlings D, Switzer L, Findlay B, Knights S. Interactive computer play as "motor therapy" for individuals with cerebral palsy. Semin Pediatr Neurol. 2013 Jun;20(2):127-38. doi: 10.1016/j.spen.2013.06.003. PMID 23948687
- [Background] Bilde PE, Kliim-Due M, Rasmussen B, Petersen LZ, Petersen TH, Nielsen JB. Individualized, home-based interactive training of cerebral palsy children delivered through the Internet. BMC Neurol. 2011 Mar 9;11:32. doi: 10.1186/1471-2377-11-32. PMID 21392370
- [Background] Fluet GG, Qiu Q, Kelly D, Parikh HD, Ramirez D, Saleh S, Adamovich SV. Interfacing a haptic robotic system with complex virtual environments to treat impaired upper extremity motor function in children with cerebral palsy. Dev Neurorehabil. 2010;13(5):335-45. doi: 10.3109/17518423.2010.501362. PMID 20828330
- [Background] Howcroft J, Klejman S, Fehlings D, Wright V, Zabjek K, Andrysek J, Biddiss E. Active video game play in children with cerebral palsy: potential for physical activity promotion and rehabilitation therapies. Arch Phys Med Rehabil. 2012 Aug;93(8):1448-56. doi: 10.1016/j.apmr.2012.02.033. Epub 2012 May 7. PMID 22571917
- [Background] Jannink MJ, van der Wilden GJ, Navis DW, Visser G, Gussinklo J, Ijzerman M. A low-cost video game applied for training of upper extremity function in children with cerebral palsy: a pilot study. Cyberpsychol Behav. 2008 Feb;11(1):27-32. doi: 10.1089/cpb.2007.0014. PMID 18275309
- [Background] Ritterband-Rosenbaum A, Christensen MS, Nielsen JB. Twenty weeks of computer-training improves sense of agency in children with spastic cerebral palsy. Res Dev Disabil. 2012 Jul-Aug;33(4):1227-34. doi: 10.1016/j.ridd.2012.02.019. Epub 2012 Mar 22. PMID 22502849
- [Background] Rostami HR, Arastoo AA, Nejad SJ, Mahany MK, Malamiri RA, Goharpey S. Effects of modified constraint-induced movement therapy in virtual environment on upper-limb function in children with spastic hemiparetic cerebral palsy: a randomised controlled trial. NeuroRehabilitation. 2012;31(4):357-65. doi: 10.3233/NRE-2012-00804. PMID 23232158
- [Background] Sandlund M, Waterworth EL, Hager C. Using motion interactive games to promote physical activity and enhance motor performance in children with cerebral palsy. Dev Neurorehabil. 2011;14(1):15-21. doi: 10.3109/17518423.2010.533329. PMID 21241174
- [Background] Sharan D, Ajeesh PS, Rameshkumar R, Mathankumar M, Paulina RJ, Manjula M. Virtual reality based therapy for post operative rehabilitation of children with cerebral palsy. Work. 2012;41 Suppl 1:3612-5. doi: 10.3233/WOR-2012-0667-3612. PMID 22317271
- [Background] Weightman A, Preston N, Levesley M, Holt R, Mon-Williams M, Clarke M, Cozens AJ, Bhakta B. Home based computer-assisted upper limb exercise for young children with cerebral palsy: a feasibility study investigating impact on motor control and functional outcome. J Rehabil Med. 2011 Mar;43(4):359-63. doi: 10.2340/16501977-0679. PMID 21347508
- [Background] Hung JW, Chou CX, Hsieh YW, Wu WC, Yu MY, Chen PC, Chang HF, Ding SE. Randomized comparison trial of balance training by using exergaming and conventional weight-shift therapy in patients with chronic stroke. Arch Phys Med Rehabil. 2014 Sep;95(9):1629-37. doi: 10.1016/j.apmr.2014.04.029. Epub 2014 May 23. PMID 24862764
- [Background] Luna-Oliva L, Ortiz-Gutierrez RM, Cano-de la Cuerda R, Piedrola RM, Alguacil-Diego IM, Sanchez-Camarero C, Martinez Culebras Mdel C. Kinect Xbox 360 as a therapeutic modality for children with cerebral palsy in a school environment: a preliminary study. NeuroRehabilitation. 2013;33(4):513-21. doi: 10.3233/NRE-131001. PMID 24018364
- [Background] Dinomais M, Veaux F, Yamaguchi T, Richard P, Richard I, Nguyen S. A new virtual reality tool for unilateral cerebral palsy rehabilitation: two single-case studies. Dev Neurorehabil. 2013 Dec;16(6):418-22. doi: 10.3109/17518423.2013.778347. Epub 2013 Jul 11. PMID 23845037
- [Background] Chang YJ, Chen SF, Huang JD. A Kinect-based system for physical rehabilitation: a pilot study for young adults with motor disabilities. Res Dev Disabil. 2011 Nov-Dec;32(6):2566-70. doi: 10.1016/j.ridd.2011.07.002. Epub 2011 Jul 23. PMID 21784612
- [Background] Randall M, Carlin JB, Chondros P, Reddihough D. Reliability of the Melbourne assessment of unilateral upper limb function. Dev Med Child Neurol. 2001 Nov;43(11):761-7. doi: 10.1017/s0012162201001396. PMID 11730151
- [Background] Thorley M, Lannin N, Cusick A, Novak I, Boyd R. Construct validity of the Quality of Upper Extremity Skills Test for children with cerebral palsy. Dev Med Child Neurol. 2012 Nov;54(11):1037-43. doi: 10.1111/j.1469-8749.2012.04368.x. Epub 2012 Jul 31. PMID 22845645
- [Background] Thorley M, Lannin N, Cusick A, Novak I, Boyd R. Reliability of the quality of upper extremity skills test for children with cerebral palsy aged 2 to 12 years. Phys Occup Ther Pediatr. 2012 Feb;32(1):4-21. doi: 10.3109/01942638.2011.602389. Epub 2011 Aug 15. PMID 21838618
- [Background] Arnould C, Penta M, Renders A, Thonnard JL. ABILHAND-Kids: a measure of manual ability in children with cerebral palsy. Neurology. 2004 Sep 28;63(6):1045-52. doi: 10.1212/01.wnl.0000138423.77640.37. PMID 15452296
- [Background] Gordon AM, Schneider JA, Chinnan A, Charles JR. Efficacy of a hand-arm bimanual intensive therapy (HABIT) in children with hemiplegic cerebral palsy: a randomized control trial. Dev Med Child Neurol. 2007 Nov;49(11):830-8. doi: 10.1111/j.1469-8749.2007.00830.x. PMID 17979861
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Jongbloed-Pereboom M, Nijhuis-van der Sanden MW, Steenbergen B. Norm scores of the box and block test for children ages 3-10 years. Am J Occup Ther. 2013 May-Jun;67(3):312-8. doi: 10.5014/ajot.2013.006643. PMID 23597689
- [Background] Wang HY, Cheng CC, Hung JW, Ju YH, Lin JH, Lo SK. Validating the Cerebral Palsy Quality of Life for Children (CP QOL-Child) questionnaire for use in Chinese populations. Neuropsychol Rehabil. 2010 Dec;20(6):883-98. doi: 10.1080/09602011.2010.509190. Epub 2010 Sep 1. PMID 20859827
- [Background] Blanche EI. Play in Occupational Therapy for Children. In: Parham LD, Fazio LS, eds. Play in children with cerebral palsy: Doing with-not doing to. 2 ed: Mosby Elsevier; 2008.
- [Background] Reid D, Campbell K. The use of virtual reality with children with cerebral palsy: A pilot randomized trial. Therapeutic Recreation Journal. 2006;40(4):255-268.
- [Background] Randall M, Johnson L, Reddihough D. The Melbourne Assessment of Unilateral Upper Limb Function: Test Administration Manual. Royal Children's Hospital - Melbourne; 1999.
- [Background] Hislop HJ, Montgomery J. Daniels and Worthingham's Muscle Testing: Techniques of Manual Examination. Elsevier Science Health Science Division; 2007.
- [Background] DeMatteo C, Law M, Russell D, Pollock N, Rosenbaum P, Walter S. QUEST: Quality of Upper Extremity Skills Test. CanChild Centre for Childhood Disability Research; 1992.
- [Background] DeMatteo C, Law M, Russell D, Pollock N, Rosenbaum P, Walter S. The Reliability and Validity of the Quality of Upper Extremity Skills Test. Physical & occupational therapy in pediatrics. 1993;13(2):1-18.
- [Background] Martin NA. Test of Visual Perceptual Skills-3. 3rd ed.: Novato, CA: American Therapy Publications; 2006.